CLINICAL TRIAL: NCT03616782
Title: Multicenter Phase II Study of Ixazomib Maintenance in Patients With Newly Diagnosed Mantle Cell Lymphoma
Brief Title: Ixazomib Maintenance in Patients With Newly Diagnosed Mantle Cell Lymphoma(MCL)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ho Sup Lee (Other)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor-Investigator, Ho Sup Lee, Professor, Kosin University Gospel Hospital
Organization: Kosin University Gospel Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FIXATION
Record Dates: First submitted 2018-07-09; First posted 2018-08-06 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — ixazomib

STUDY DESIGN:
Intervention Model Description: Ixazomib 3mg on day 1, 8, 15 q 4 weeks for 24months or untile to progression
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ixazomib (Experimental): Ixazomib 3mg on day a, 8, 15 q 4 weeks for 24 months or until to progression
  Interventions: Drug: Ixazomib

INTERVENTIONS:
Drug: Ixazomib — Ixazomib 3mg on day 1, 8, 15 q 4 weeks for 24 months or until progression

SUMMARY:
1. Induction chemotherapy 1) RCHOP(Rituximab+Cyclophosphamide+Doxorubicin+Vincristine+Prednisone) 2) VR-CAP (Bortezomib+Rituximab+Cyclophosphamide+Doxorubicin+Prednisone)

   Patients who have received induction chemotherapy will be evaluated for responses and those who achieved more than PR(Partial response) or PR will be eligible for this study after receiving informed consents.
2. Experimental step Maintenance ixazomib beginning at least 8 weeks after completion of induction chemotherapy, patients receive ixazomib per oral 3 mg on day 1, 8, and 15 for 4 weeks. And the dose of ixazomib can be escalated to 4mg by response such as partial response or MRD positive. Treatment repeats every 4 weeks for up to 24 months in the absence of disease progression or unacceptable toxicity.

Patients are screened and sign the informed consent after completion induction chemotherapy (RCHOP or VR-CAP) with more than PR or PR confirmed. It is likely to take approximately 8 weeks in performing above procedures.

Patients start maintenance therapy at least 8 weeks and also can be allowed for the extension of 4 weeks because of delayed response evaluation, recovery toxicities of chemotherapy, and official process including agree with informed consent. Recently, ongoing studies about maintenance therapy in lymphoma have window periods of 8-12 weeks.

Ixazomib maintenance should continue for 2 years.

DETAILED DESCRIPTION:
1. Induction chemotherapy 1) RCHOP: Before enrollments, patients receive comprising R-CHOP, as induction therapy, comprised rituximab (at a dose of 375 mg per square meter of body-surface area), cyclophosphamide (750 mg per square meter), doxorubicin (50 mg per square meter), vincristine (1.4mg per square meter) administered on days 1, and oral prednisone (100 mg per square meter) administered on days 1 to 5. Patients also receive pegylated granulocyte-colonly stimulating factor (G-CSF) subcutaneously (SC) on day 2 to day 5. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

   VR-CAP: Before enrollments, patients receive comprising VR-CAP, as induction therapy, comprised bortezomib (1.3 mg per square meter of body-surface area) administered on days 1, 4, 8, 11, rituximab (at a dose of 375 mg per square meter), cyclophosphamide (750 mg per square meter), doxorubicin (50 mg per square meter) administered on days 1, and oral prednisone (100 mg per square meter) administered on days 1 to 5. Patients also receive pegylated G-CSF SC on day 2 to day 5. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

   Patients who have received induction chemotherapy will be evaluated for responses and those who achieved more than PR(Partial response) or PR will be eligible for this study after receiving informed consents.
2. Experimental step Maintenance ixazomib beginning at least 8 weeks after completion of induction chemotherapy, patients receive ixazomib per oral 3 mg on day 1, 8, and 15 for 4 weeks. And the dose of ixazomib can be escalated to 4mg by response such as partial response or MTD(Maximum Tolerated Dose) positive. Treatment repeats every 4 weeks for up to 24 months in the absence of disease progression or unacceptable toxicity.

Patients are screened and sign the informed consent after completion induction chemotherapy (RCHOP or VR-CAP) with more than PR or PR confirmed. It is likely to take approximately 8 weeks in performing above procedures.

Patients start maintenance therapy at least 8 weeks and also can be allowed for the extension of 4 weeks because of delayed response evaluation, recovery toxicities of chemotherapy, and official process including agree with informed consent. Recently, ongoing studies about maintenance therapy in lymphoma have window periods of 8-12 weeks.

Ixazomib maintenance should continue for 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged ≥19 years
2. Histologically confirmed mantle cell lymphoma (MCL) meeting the following criteria: determined by histology and either expression of cyclin D1 (in association with CD20 and CD5) or evidence of t(11;14) translocation (by cytogenetics, fluorescence in-situ hybridization, or polymerase chain reaction)
3. In all patients, a paraffin-embedded biopsy tissue block or slides (preferably of lymph node origin or bone marrow) was sent to central laboratories (Diagnostic Cytology Laboratories or department of pathology) for confirmation of diagnosis of MCL.
4. Stage II, III, or IV
5. Patients who received RCHOP or VR-CAP induction chemotherapy for 6 cycles confirmed response as more than PR or PR after induction therapy and who are ineligible for transplantation. .
6. No clinical evidence of central nervous system (CNS) involvement by lymphoma
7. Patients must have measurable disease; CT scans at baseline are required to define the extent of measurable disease; the scans must be obtained within 6 weeks prior to registration; combined CT/PET scans may be used for the baseline and subsequent evaluations if accurate tumor measurements can be obtained from the CT component
8. Eastern Cooperative Oncology Group (ECOG) performance status 0-2
9. Absolute neutrophil count (ANC) > 1,000 mm^3 (unless low count due to marrow involvement or splenomegaly)
10. Platelets > 75,000 mm^3 (unless low counts due to marrow involvement or splenomegaly)
11. Creatinine clearance of ≥ 30 mL/min
12. Total bilirubin ≤ 1.5 x the upper limit of normal (may be up to 3.0 mg/dL if due to Gilbert's disease or due to liver involvement by lymphoma), alanine transaminase level ≤3 times the upper limit of normal; aspartate transaminase level ≤3 times the upper limit of normal
13. Patients over the age of 45 must have a left ventricular ejection fraction (LVEF) of greater than 45% documented within 90 days prior to registration
14. Female patients had to be post-menopausal for ≥1 year, surgically sterile, or practicing an effective method of birth control (as described in the protocol), and have a negative serum beta-human chorionic gonadotropin or urine pregnancy test at screening; they also had to agree to continue using birth control measures for ≥6 months after terminating treatment. Male patients had to agree to use an acceptable method of contraception for the duration of the study.

Exclusion Criteria:

1. Female patients who are lactating or have a positive serum pregnancy test during the screening period.
2. Grade 2 or higher baseline peripheral neuropathy
3. Major surgery within 14 days before enrollment.
4. Radiotherapy within 14 days before enrollment. If the involved field is small, 7 days will be considered a sufficient interval between treatment and administration of the ixazomib.
5. Central nervous system involvement.
6. Infection requiring systemic antibiotic therapy or other serious infection within 14 days before study enrollment.
7. Evidence of current uncontrolled cardiovascular conditions, including uncontrolled hypertension, uncontrolled cardiac arrhythmias, symptomatic congestive heart failure, unstable angina, or myocardial infarction within the past 6 months.
8. Systemic treatment, within 14 days before the first dose of ixazomib, with strong CYP3A inducers (rifampin, rifapentine, rifabutin, carbamazepine, phenytoin, phenobarbital), or use of St. John's wort.
9. Active systemic infection requiring treatment, a known diagnosis of human HIV, or active hepatitis B (hepatitis B carriers were permitted)
10. Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol.
11. Known allergy to any of the study medications, their analogues, or excipients in the various formulations of any agent.
12. Known gastrointestinal(GI) disease or GI procedure that could interfere with the oral absorption or tolerance of ixazomib including difficulty swallowing.
13. Diagnosed or treated for another malignancy within 2 years before study enrollment or previously diagnosed with another malignancy and have any evidence of residual disease. Patients with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection.
14. Patient has more than Grade 2 peripheral neuropathy on clinical examination during the screening period.
15. Participation in other clinical trials, including those with other investigational agents not included in this trial, within 30 days of the start of this trial and throughout the duration of this trial.
16. Patients that have previously been treated with ixazomib, or participated in a study with ixazomib whether treated with ixazomib or not.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2018-12-24 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
2-year PFS rates in adult patients with newly diagnosed Mantle Cell Lymphoma | 2years

SECONDARY OUTCOMES:
Complete Response (CR) achievement rates after ixazomib maintenance by Lugano classification | an average of 2 year
Overall survival (OS) rates at 2 years | 2years
  overall survival of patients with Mantle Cell Lymphoma
Adverse events (AEs) | 2years
  Adverse events will be measured by the CTCAE scale, version 4.03
Time to relapse/progression | 2years
  Time to progression is measured from the date of start of study to the date of relapse/progression
Time to next therapy (TTNT) | 2years
Minimal residual disease (MRD) by IgH or IgK NGS from BM, lymphoma tissue at the baseline and then peripheral blood (cell free DNA). | Screening, 24weeks, 4weeks after end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Ho Sup Lee, MD, Principal Investigator — Kosin University Gospel Hospital
Locations (1):
- Kosin University Gospel Hospital, Busan, Western, South Korea